CLINICAL TRIAL: NCT05822921
Title: Providing Accessible Diagnostic Evaluations and Psychoeducation for Autism Spectrum Disorder in Rural Southwest Virginia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: Autism Speaks (Other); University of Virginia (Other); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-423; UL1TR003015 (NIH)
Record Dates: First submitted 2023-02-01; First posted 2023-04-21 (Actual); Results first posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-10

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Parents of children who meet criteria for a diagnosis of autism spectrum disorder (ASD) will be randomized into one of three groups (i.e., in-person psychoeducation, telehealth psychoeducation, or "psychoeducation as usual" with paper psychoeducation materials).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- In-person Psychoeducation (Experimental)
  Interventions: Behavioral: In-person Psychoeducation (IP)
- Telehealth Psychoeducation (Experimental)
  Interventions: Behavioral: Telehealth Psychoeducation (TH)
- Psychoeducation as Usual (Active Comparator)
  Interventions: Behavioral: Psychoeducation as Usual (PAU)

INTERVENTIONS:
Behavioral: In-person Psychoeducation (IP) — Parents will attend two 60-minute (i.e. one day per week, for the next two weeks), in-person psychoeducation sessions on the MAC, in or near their hometown. During these sessions, a clinician will discuss a series of psychoeducation topics supplemented with PowerPoint slides. Across the two sessions, the following topics will be covered: (1) signs/symptoms and epidemiology of ASD, (2) risk factors associated with developing ASD (e.g., genetics, neurobiology, environment, social motivation), (3) navigating the IEP process, and (4) evidence-based best practices recommended for their child's profile of ASD symptoms and co-occurring conditions. This delivery method will allow parents to ask questions and receive immediate, live, and detailed answers from an expert clinician, to focus on specific examples relevant to their child, and to foster ASD knowledge and efficacy in helping their child.
  Arms: In-person Psychoeducation
Behavioral: Telehealth Psychoeducation (TH) — Parents in this group will attend two 60-minute sessions, remotely via a live video chat platform, rather than in-person. Otherwise, it will follow the same format and PowerPoint materials as the IP Group. Sessions will still be facilitated by a clinician, thus maintaining the option to ask questions, discuss personalized examples, etc. For families without computer and internet access, the family will be assisted with to connecting to internet access at a private and convenient location (e.g., a church, library, or local community services agency). In the event that this is not possible, the family will be randomized to one of the other two groups.
  Arms: Telehealth Psychoeducation
Behavioral: Psychoeducation as Usual (PAU) — Parents in this group will receive basic paper psychoeducation resources, distributed at their feedback session. It will be up to each parent how frequently and diligently these resources are reviewed. This should be akin to what a family might have access to at their pediatric or primary care office. To be consistent across study groups, the materials produced for these parents will be comprehensive and will include the same span of content as the PowerPoint slides used in the other two groups, but without structured sessions facilitated by a clinician. Upon distribution of materials, parents will be provided with our contact information and encouraged to reach out if any questions occur. Parents in the paper informational materials group will have the option to complete two in-person or video conference psychoeducation sessions after the end of the study, if preferred (i.e., 6 months later).
  Arms: Psychoeducation as Usual

SUMMARY:
This study will be the pilot/feasibility phase of a future clinical trial. The proposed feasibility and pilot study aims to bridge the barriers to diagnosis by providing easy-to-access assessment for free, through a mobile unit that travels to rural locations and telehealth assessments. The diagnostic evaluation will confirm or rule out a diagnosis of ASD, followed by purposeful ASD psychoeducation for parents whose children are diagnosed.

Parents of children who meet criteria for a diagnosis of autism spectrum disorder (ASD) or are suspected to have ASD will be randomized into one of three groups (i.e., in-person psychoeducation, telehealth psychoeducation, or "psychoeducation as usual" with paper psychoeducation materials). Parents will complete outcome measures related to their satisfaction, empowerment, and autism spectrum disorder knowledge. Changes in empowerment and ASD knowledge from pre- to post- psychoeducation will be measured using t-tests. The investigators will also track if participants sought and/or received additional ASD-related services throughout the study up to 6-months post-psychoeducation. Results from this study will help to guide a future, fully powered efficacy trial with a larger sample.

Added April 2020: In light of the Virginia governor's stay-at-home order in response to the COVID-19 outbreak, the investigators are altering the protocol in line with the university's request to move to remote conduct of research where possible as well as to continue to provide services to families in this time, in line with Executive Order 53 from the VA Governor. Parents in the latter half of the study conducted entirely remotely, will be randomized into the two psychoeducation conditions, telehealth or paper materials psychoeducation groups, as in-person visits are not permitted. Statistical analyses will be added to compare results between and within those who received in-person versus telehealth assessments. The investigators and participants may return to in-person assessments if and when it is possible to do so, but reserve the right to continue tele-assessment even once stay-at-home orders are lifted, in order to fully answer the research aim of the feasibility and validity or tele-assessment procedures in ASD.

DETAILED DESCRIPTION:
This study will be the pilot/feasibility phase of a future clinical trial. The proposed feasibility and pilot study aims to bridge the barriers to diagnosis by providing easy-to-access assessment for free, through a mobile unit that travels to rural locations and telehealth assessments. The diagnostic evaluation will confirm or rule out a diagnosis of ASD, followed by purposeful ASD psychoeducation for parents whose children are diagnosed.

Parents of children who meet criteria for a diagnosis of autism spectrum disorder (ASD) or are suspected to have ASD will be randomized into one of three groups (i.e., in-person psychoeducation, telehealth psychoeducation, or "psychoeducation as usual" with paper psychoeducation materials). Parents will complete outcome measures related to their satisfaction, empowerment, and autism spectrum disorder knowledge. Changes in empowerment and ASD knowledge from pre- to post-psychoeducation will be measured using t-tests. The investigators will also track if participants sought and/or received additional ASD-related services throughout the study, up to 6-months post-psychoeducation. Results from this study will help to guide a future, fully powered efficacy trial with a larger sample.

Added April 2020:

In light of the Virginia governor's stay-at-home order in response to the COVID-19 outbreak, which reached pandemic status approximately halfway through data collection, all in-person research and clinical services have been paused at Virginia Tech as of March 13, 2020. To continue to provide services to families in this time, in line with Executive Order 53 from the VA Governor to ensure that the stay-at-home orders do not limit the provision of health care or medical services, this study will begin exploring the feasibility of conducting tele-assessment, a comprehensive assessment battery via a secure video platform and phone.

As such, the protocol is altered to be in line with the university's request to move to remote conduct of research where possible. For the remaining half of participants, the investigators will replace the mobile assessment battery with a tele-assessment battery, delivered via secure online video platform ZoomHIPAA and/or by phone (totaling up to 7 hours of assessment). As such, the protocol is revised to include tele-assessments (no in-person assessments) and randomly assigning eligible participants to either the telehealth or paper materials psychoeducation groups. All outcome measures will remain the same, but will be collected online or by telephone. The investigators and participants may return to in-person assessments if and when it is possible, but reserve the right to continue tele-assessment even once stay-at-home orders are lifted.

The aims of the project will be altered somewhat by the updated procedure. The study will be significantly underpowered to analyze the differences between psychoeducation conditions within and between each assessment modality (i.e., in-person vs. telehealth), therefore in person and telehealth conditions will be combined into one psychoeducation (PE) group with clinician-led sessions. The mean differences between the PE group and the psychoeducation as usual (i.e., paper materials) formats will be preliminarily explored, in terms of both feasibility and satisfaction of the psychoeducation services and changes in outcome measures (i.e., FES and ASK-Q). Pending permission to return to in-person assessments, analyses will also report alignment between diagnoses made via tele-assessment (CARS-2 and ADI-R) and a later in-person administration of the ADOS-2.

ELIGIBILITY:
Inclusion Criteria:

* Parent(s)/Caregiver(s) to a child between the ages of 16 months through 17 years old with autism concern, who are seeking a diagnostic assessment, and live in a rural underserved community
* Recruitment in line with gender ratio seen in the prevalence of ASD (i.e., 4.2 boys to 1 girl)
* English-speaking parent
* Added April 2020: For the second half of the study (Tele-assessment), parents must have a computer, laptop, or tablet (at least 9.7 inches diagonally) with web-camera and stable Internet.

Exclusion Criteria:

* Children participants who will turn 18 before their participation in the study has ended
* If a family does not have Internet and computer access, the family will not be excluded, but will be randomized into a group other than the telehealth psychoeducation group.

Ages: 16 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2021-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Scarpa, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (2):
- United States (2):
  - Virginia Tech, Blacksburg, Virginia
  - Mount Rogers Community Services, Wytheville, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The # of participants completing the study refer to child-parent pairs rather than individuals. A diagnostic evaluation for autism spectrum disorder was conducted for the child. One child did not meet ASD criteria, so that family was not assigned, leaving a final total of 20 parent-child pairs. Due to COVID-19, the protocol was revised such that participants who received either telehealth or in-person psychoeducation were grouped in a single arm (i.e., Psycho-education Clinician-led).
Groups:
- Psychoeducation (PE) Clinician-led Sessions: Parents will attend two 60-minute psychoeducation sessions (either in person or via Zoom). During these sessions, a clinician will discuss a series of psychoeducation topics supplemented with PowerPoint slides. Across the two sessions, the following topics will be covered: (1) signs/symptoms and epidemiology of ASD, (2) risk factors associated with developing ASD (e.g., genetics, neurobiology, environment, social motivation), (3) navigating the IEP process, and (4) evidence-based best practices recommended for their child's profile of ASD symptoms and co-occurring conditions. This delivery method will allow parents to ask questions and receive immediate, live, and detailed answers from an expert clinician, to focus on specific examples relevant to their child, and to foster ASD knowledge and efficacy in helping their child.
- Psychoeducation as Usual (PAU): Parents in this group will receive basic paper psychoeducation resources, distributed at their feedback session. It will be up to each parent how frequently and diligently these resources are reviewed. This should be akin to what a family might have access to at their pediatric or primary care office. To be consistent across study groups, the materials produced for these parents will be comprehensive and will include the same span of content as the PowerPoint slides used in the other two groups, but without structured sessions facilitated by a clinician. Upon distribution of materials, parents will be provided with our contact information and encouraged to reach out if any questions occur.
Period: Overall Study
Arm/Group | Psychoeducation (PE) Clinician-led Sessions | Psychoeducation as Usual (PAU)
Started | 11 | 9
Completed | 10 | 8
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: Numbers refer to parent-child pairs, not individual participants. That is, 11 parent-child pairs completed the PE arm and 9 parent-child pairs completed the PAU arm. Baseline characteristics of age, sex, race, ethnicity, and region are reported for the children. Age, sex, and region are also reported for the parents. Reference to either parents or children is specified in the measure description.
Groups:
- Total: Total of all reporting groups
Arm/Group | Psychoeducation (PE) Clinician-led Sessions | Psychoeducation as Usual (PAU) | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Categorical [Count of Participants; unit: Participants] — For children
  Participants
    <=18 years | 11 | 9 | 20
    Between 18 and 65 years | 0 | 0 | 0
    >=65 years | 0 | 0 | 0
Age, Categorical [Count of Participants; unit: Participants] — For parents
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 11 | 9 | 20
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] — For children
  years | 5.91 [2 to 10] | 8.78 [2 to 14] | 7.2 [2 to 14]
Age, Continuous [Mean (Full Range); unit: years] — For parents
  years | 34.55 [24 to 47] | 34.56 [25 to 45] | 34.55 [24 to 47]
Sex: Female, Male [Count of Participants; unit: Participants] — For children
  Participants
    Female | 5 | 1 | 6
    Male | 6 | 8 | 14
Sex: Female, Male [Count of Participants; unit: Participants] — For parents
  Participants
    Female | 10 | 8 | 18
    Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — For children
  Participants
    Hispanic or Latino | 0 | 0 | 0
    Not Hispanic or Latino | 11 | 9 | 20
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — For children
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 3 | 3
    White | 10 | 5 | 15
    More than one race | 1 | 1 | 2
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — For children
  participants
    United States | 11 | 9 | 20
Region of Enrollment [Number; unit: participants] — For parents
  participants
    United States | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Parent-child Pairs Who Completed Study Sessions Assessed by Parental Attendance
Description: Retention of participants assessed by parental attendance for all study sessions. Only parental attendance to psycho-education sessions was included for this measure. Child attendance was not needed.
Time Frame: Time 1: Baseline/intake (0 weeks); Time 2: Pre-intervention (2 weeks); Time 3: Immediately post-intervention (4 weeks after baseline); Time 4: 6- week followup (10 weeks after baseline); Time 5: 6-month followup (7 months after baseline)
Population: Number of child-parent pairs enrolled in the study and randomized to each condition. For the PE condition, two families were in person and nine families had sessions conducted over Zoom. For the PAU condition, all families received paper materials.
Measure: Number; unit: parent-child pairs
Arm/Group | Psychoeducation (PE) Clinician-led Sessions | Psychoeducation as Usual (PAU)
Number analyzed (Participants) | 11 | 9
parent-child pairs
  Time 1: Baseline/Intake into arms (0 weeks) | 11 | 9
  Time 2: Pre-intervention (2 weeks) | 11 | 9
  Time 3: Immediately Post-intervention (4 weeks after baseline) | 10 | 8
  Time 4: 6-week follow-up (10 weeks after baseline) | 7 | 5
  Time 5: 6-month follow-up (7 months after baseline) | 9 | 6

2. Primary Outcome: Parent Satisfaction Assessed Via SATISFACTION SURVEY
Description: SATISFACTION SURVEY: A satisfaction survey will be administered to elicit parents' feedback on our service.Satisfaction survey administered immediately post-psychoeducation, on a scale of 0=completely disagree to 4= completely agree with statements about satisfaction with psychoeducation received, ability to function day to day, learning throughout materials, ability to handle situations with child in future, and ability to gain a better outlook on life with child. Total sum scores were used, for a range of 0 to 20, with higher scores indicating greater satisfaction.
Time Frame: immediately post-intervention (4 weeks after baseline)
Population: For the PE condition, two families were in person and nine families had sessions conducted over Zoom. For the PAU condition, all families received paper materials. One family in each condition did not complete the post-intervention measures, leaving 10 in the PE condition and 8 in the PAU condition. All measures were completed by parents in the parent-child pair. Outcome measures were not collected from children.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Psychoeducation (PE) Clinician-led Sessions | Psychoeducation as Usual (PAU)
Number analyzed (Participants) | 10 | 8
score on a scale | 19.5 [17 to 20] | 17.38 [10 to 20]
Statistical Analysis 1: Comparison: Psychoeducation (PE) Clinician-led Sessions vs Psychoeducation as Usual (PAU); Test type: Other — Independent t-test was used; p = .871, t-test, 2 sided

3. Secondary Outcome: Change in Parental Empowerment Assessed by the FAMILY EMPOWERMENT SCALE
Description: Parental empowerment will be assessed by the Family Empowerment Scale and compared across education delivery formats. The Family Empowerment Scale measures levels of perceived efficacy in community involvement, navigating services for child and family. This scale includes three areas (family domain, service system domain, and community/political domain). Range of scores per domain include: family domain (12 to 60), service system domain (12 to 60), and community/political domain (10 to 50). Total sum scores could range from 34 - 170. A higher score indicates greater empowerment in a given domain. Change in sum total score across all domains from pre- to post-psychoeducation was used for analysis.
Time Frame: 2 weeks from start of study (pre-psychoeducation) to 4 weeks from start of study (post-psychoeducation)
Population: Families who completed each arm were included in the analyses. One family in each arm did not complete the measures at post-intervention. All measures were completed by parents in the parent-child pair. Outcome measures were not collected from children.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psychoeducation (PE) Clinician-led Sessions | Psychoeducation as Usual (PAU)
Number analyzed (Participants) | 10 | 8
units on a scale | 7 (8.35) | 7.88 (18.81)
Statistical Analysis 1: Comparison: Psychoeducation (PE) Clinician-led Sessions vs Psychoeducation as Usual (PAU); Test type: Other — Independent t-test was used; p = 0.896, t-test, 2 sided

4. Secondary Outcome: Change in Parental Knowledge Assessed by AUTISM STIGMA AND KNOWLEDGE QUESTIONNAIRE
Description: Parental knowledge will be assessed using the AUTISM STIGMA AND KNOWLEDGE QUESTIONNAIRE. Total sum scores range from minimum score = 0 to maximum score = 48. A higher raw score is better and indicates more autism knowledge and less autism stigma. Change score from pre- to post- psychoeducation was used for analysis.
Time Frame: 2 weeks from start of study (pre-psychoeducation) to 4 weeks from start of study (post-psychoeducation)
Population: Families in both arms who completed psycho-education were included in analyses. One family in each arm did not complete the post-intervention measures. All measures were completed by parents in the parent-child pair. Outcome measures were not collected from children.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psychoeducation (PE) Clinician-led Sessions | Psychoeducation as Usual (PAU)
Number analyzed (Participants) | 10 | 8
units on a scale | 1.4 (1.43) | 0.5 (2.507)
Statistical Analysis 1: Comparison: Psychoeducation (PE) Clinician-led Sessions vs Psychoeducation as Usual (PAU); Test type: Other — Independent t-test was used; p = 0.351, t-test, 2 sided

5. Secondary Outcome: Use of Additional Autism Spectrum Disorder-related Services Assessed by NEW SERVICES SURVEY
Description: Use of additional Autism Spectrum Disorder-related services accessed will be assessed using a NEW SERVICES SURVEY. Parents will be surveyed as to what new services have been used since the last session or survey time point. This survey will ask whether parents have contacted other service agencies, the date of contact, whether they received any new services (and to specify the services received), and the date of first service received.
Time Frame: Time 2: pre-intervention (2 weeks after baseline), Time 3: immediately post-intervention (4 weeks after baseline), Time 4: 6-week followup (10 weeks after baseline), to Time 5: 6-month followup (7 months after baseline)
Population: Percentage of families who received any additional services from the prior time-point at any point after the psycho-education, from pre-intervention (2 weeks after baseline) up to 6 month followup (7 months after baseline). All measures were completed by parents in the parent-child pair. Outcome measures were not collected from children.
Measure: Number; unit: percentage of families
Arm/Group | Psychoeducation (PE) Clinician-led Sessions | Psychoeducation as Usual (PAU)
Number analyzed (Participants) | 11 | 9
percentage of families | 81.83 | 55.56

ADVERSE EVENTS:
Description: Death, serious adverse events, and other (non-serious adverse events) were not assessed for this study.
Arm/Group | Psychoeducation (PE) Clinician-led Sessions | Psychoeducation as Usual (PAU)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Small sample size. In person and Zoom psychoeducation sessions were combined into one arm because COVID-19 pandemic necessitated a pivot to Zoom. As such, we had only completed 2 in person sessions before shifting to all Zoom sessions. Additionally, while 20 families were randomized to conditions, only 18 completed the post-psychoeducation measures, and only 15 completed the 6-month follow-up measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-18): https://cdn.clinicaltrials.gov/large-docs/21/NCT05822921/Prot_SAP_000.pdf